CLINICAL TRIAL: NCT07288359
Title: An Open-label, Multi-center, Phase I/II Study of GVV858 as a Single Agent and in Combination With Endocrine Therapy in Patients With Advanced Hormone Receptor Positive, HER2- Negative Breast Cancer and Other Advanced Solid Tumors
Brief Title: Study of GVV858 as a Single Agent or in Combination With Endocrine Therapy in Patients With HR+/HER2- Breast Cancer and Other Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CGVV858A12101; 2025-521911-38 (Other: CTIS)
Record Dates: First submitted 2025-12-15; First posted 2025-12-17 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Advanced HR+/HER2- Breast Cancer; Advanced CCNE1-amplified Solid Tumors; Metastatic Castration-resistant Prostate Cancer
Keywords: GVV858; Fulvestrant; Letrozole; Breast Cancer; CCNE1 amplification; Prostate Cancer
MeSH Terms: conditions — Breast Neoplasms; Prostatic Neoplasms | interventions — Fulvestrant; Letrozole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- GVV858 Single Agent (Arm A) (Experimental): Phase I
  Interventions: Drug: GVV858
- GVV858 in combination with fulvestrant (Arm B) (Experimental): Phase I
  Interventions: Drug: GVV858; Drug: Fulvestrant
- GVV858 in combination with letrozole (Arm C) (Experimental): Phase I
  Interventions: Drug: GVV858; Drug: Letrozole
- GVV858 in combination with fulvestrant (Arm D) (Experimental): Phase II, recommended dose regimen 1
  Interventions: Drug: GVV858; Drug: Fulvestrant
- GVV858 in combination with fulvestrant (Arm E) (Experimental): Phase II, recommended dose regimen 2, optional dose optimization
  Interventions: Drug: GVV858; Drug: Fulvestrant

INTERVENTIONS:
Drug: GVV858 — Experimental
Drug: Fulvestrant — Approved medication
  Other Names: Faslodex
  Arms: GVV858 in combination with fulvestrant (Arm B); GVV858 in combination with fulvestrant (Arm D); GVV858 in combination with fulvestrant (Arm E)
Drug: Letrozole — Approved medication
  Other Names: Femara
  Arms: GVV858 in combination with letrozole (Arm C)

SUMMARY:
Phase I: Characterize safety and tolerability of GVV858 as a single agent and in combination with fulvestrant or letrozole. Identify dose range for optimization/recommended dose for further clinical evaluation.

Phase II: Further characterize the safety and tolerability of GVV858 in combination with fulvestrant in patients with hormone receptor-positive/human epidermal growth factor receptor 2-negative (HR+/HER2-) advanced breast cancer.

DETAILED DESCRIPTION:
This is a first-in-human, open-label, phase I/II, multi-center study consisting of a GVV858 single agent treatment arm in patients with advanced HR+/HER2- breast cancer, other advanced solid tumors harboring CCNE1 amplification, and metastatic castration-resistant prostate cancer, and a combination treatment arm of GVV858 with fulvestrant or letrozole in patients with advanced HR+/HER2- breast cancer. Single agent escalation may be followed by an expansion part stratified by disease indication. The escalation of the fulvestrant combination arm may continue into a randomized, open label, Phase II with optional dose optimization in advanced HR+/HER2- breast cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old.
* Patients with one of the following histologically or cytologically confirmed advanced cancers:

Phase I (patients with one of the following cancers, from whom no standard therapy is available or appropriate in the judgment of the investigator):

* HR+/HER2- advanced breast cancer (aBC) with disease progression on or following at least one line of hormone-based therapy in combination with a CDK4/6i and at least one additional line of systemic therapy for metastatic disease.
* Locally advanced or metastatic cancer with a CCNE1 amplification. For dose expansion only: no more than 3 prior lines of therapy for advanced or metastatic disease.
* Metastatic castration-resistant prostate adenocarcinoma, with no documented neuroendocrine component, castrate level of testosterone, and no more than 3 prior lines of systemic therapy for metastatic disease.

Phase II:

* HR+/HER2- aBC with disease progression on or after an endocrine therapy in combination, with a CDK4/6 inhibitor for advanced disease with no more than 2 lines of endocrine therapy and no prior cytotoxic chemotherapy or antibody-drug-conjugate for advanced disease.

  - Measurable disease as determined by RECIST v1.1.
* BC only: If no measurable disease is present, then at least one predominantly lytic bone lesion must be present that can be accurately assessed at baseline and is suitable for repeated assessment.
* metastatic Castration-Resistant Prostate Cancer (mCRPC) only: If no measurable disease is present per PCWG3 modified RECIST, then at least 1 metastatic lesion must be present on bone scan imaging.

Exclusion Criteria:

* Patients with inadequate bone marrow and/or organ functions with out-of-range laboratory values.
* Clinically significant, uncontrolled heart disease and/or cardiac repolarization abnormality including myocardial infarction (MI), coronary artery bypass graft (CABG), long QT syndrome, or risk factors for Torsades de Pointes (TdP).
* Presence of symptomatic central nervous system (CNS) metastases or CNS metastases that require local therapy or increasing doses of corticosteroids within 2 weeks prior to study entry.
* Patients with symptomatic visceral disease, including visceral crisis.
* For patients with BC: Patient is concurrently using hormone replacement therapy.
* Women of childbearing potential who are unwilling to use highly effective contraception methods, pregnant or nursing women.

Other protocol-defined inclusion/exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 205 (Estimated)
Dates: Start 2025-12-29 (Actual); Primary Completion 2031-04-24 (Estimated); Study Completion 2031-05-09 (Estimated)

PRIMARY OUTCOMES:
Phase I: Incidence and severity of dose-limiting toxicities (DLTs) | 28 days
  Number of participants with DLTs. A DLT is defined as an adverse event or abnormal laboratory value of Common Terminology Criteria for Adverse Events (CTCAE) grade 3 or higher, unless clearly and inconvertibly assessed as due to disease progression, inter-current illness/injury, concomitant medications, or extraneous causes, that occurs within the first 28 days of treatment in the Phase 1 part. Other clinically significant toxicities may be considered to be DLTs, even if not CTCAE grade 3 or higher.
Phase I and phase II: Incidence and severity of adverse events (AEs) and serious adverse events (SAEs) | Up to approximately 2 years
  Number of participants with AEs and SAEs, including changes in vital signs, electrocardiograms (ECGs) and laboratory values qualifying and reported as AEs.
Phase I and phase II: Frequency of dose interruptions, reductions and discontinuations | Up to approximately 2 years
  Number of participants with dose adjustments (reductions, interruption, or permanent discontinuation) as a measure of tolerability.
Phase I and phase II: Dose intensity | Up to approximately 2 years
  The dose intensity of each study drug is computed as the ratio of actual cumulative dose received and actual duration of exposure.

SECONDARY OUTCOMES:
Phase I and II: Peak plasma concentration (Cmax) of GVV858 | Cycle 1 Day 1 and/or Day 21: From pre-dose up to maximum 24 hours post dose. The duration of one cycle is 28 days.
  Pharmacokinetic (PK) parameters calculated based on GVV858 plasma concentrations.
Phase I and II: Time to reach peak plasma concentration (Tmax) of GVV858 | Cycle 1 Day 1 and/or Day 21: From pre-dose up to maximum 24 hours post dose. The duration of one cycle is 28 days.
  PK parameters calculated based on GVV858 plasma concentrations.
Phase I and II: Area under the plasma concentration-time curve (AUC) of GVV858 | Cycle 1 Day 1 and/or Day 21: From pre-dose up to maximum 24 hours post dose. The duration of one cycle is 28 days.
  PK parameters calculated based on GVV858 plasma concentrations.
Phase I and Phase II: Overall response rate (ORR) | Up to approximately 2 years
  Tumor response assessed by the investigator based on Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v1.1), or Prostate Cancer Working Group 3 (PCWG3) criteria including PCWG3-modified RECIST v1.1. (only for patients with prostate cancer).
  ORR per RECIST v1.1 is defined as the proportion of patients with a best overall response of Complete response (CR) or Partial response (PR) according to RECIST v1.1 as per local review.
Phase I and Phase II: Best overall response (BOR) | Up to approximately 2 years
  Tumor response assessed by the investigator based on based on RECIST v1.1, or PCWG3 criteria including PCWG3-modified RECIST v1.1. (only for patients with prostate cancer).
  BOR per RECIST v1.1 is defined as the best overall confirmed response recorded from the start of the treatment until progressive disease (PD), death, start of new therapy, withdrawal of consent or end of study, whatever comes first.
Phase I and Phase II: Disease control rate (DCR) | Up to approximately 2 years
  Tumor response assessed by the investigator based on based on RECIST v1.1, or PCWG3 criteria including PCWG3-modified RECIST v1.1. (only for patients with prostate cancer).
  DCR per RECIST v1.1 is defined as the proportion of patients with a BOR of CR, PR, or Stable disease (SD) according to RECIST v1.1 as per local review.
Phase I and Phase II: Clinical benefit rate (CBR) | Up to approximately 2 years
  Tumor response assessed by the investigator based on based on RECIST v1.1, or PCWG3 criteria including PCWG3-modified RECIST v1.1. (only for patients with prostate cancer).
  CBR per RECIST v1.1 is defined as the proportion of patients with a BOR of CR, PR, or an overall lesion response of SD or Non-CR/Non-PD which lasts for at least 24 weeks according to RECIST v1.1 as per local review.
Phase I and Phase II: Progression free survival (PFS) | Up to approximately 2 years
  Tumor response assessed by the investigator based on based on RECIST v1.1, or PCWG3 criteria including PCWG3-modified RECIST v1.1. (only for patients with prostate cancer).
  PFS per RECIST 1.1 is defined as the time from the date of start of study treatment (phase I) or the date of randomization (Phase II) to the date of the first documented progression or death due to any cause.
Phase II: Duration of response (DOR) | Up to approximately 2 years
  Tumor response assessed by the investigator based on based on RECIST v1.1, or PCWG3 criteria including PCWG3-modified RECIST v1.1. (only for patients with prostate cancer).
  DOR per RECIST v1.1 is the time between the first documented response (CR or PR) and the date of progression by local review as applicable or death due to any cause.

CONTACTS AND LOCATIONS:
Locations (3):
- Tennessee Oncology PLLC, Nashville, Tennessee, United States
- Novartis Investigative Site, Singapore, Singapore
- Novartis Investigative Site, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations. This trial data availability is according to the criteria and process described on https://www.clinicalstudydatarequest.com/.